CLINICAL TRIAL: NCT04966091
Title: Working IVF Patients' Quality of Life
Acronym: WIQoL
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0426
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: In Vitro Fertilization (IVF); Infertility
Keywords: Infertility; Assisted Reproductive Techniques; quality of life; work; personal and professional interactions; depression
MeSH Terms: conditions — Infertility; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Completion of questionnaires — The quality of life questionnaire will be completed before starting the treatment and then during the embryo transfer and will be followed up at each embryo transfer over a maximum period of 18 months. We will also evaluate by means of a specific questionnaire the importance of work/life interactions management and consequences of absenteeism at work, consequences on professional evolution, anxious repercussions in the professional and private domains).

SUMMARY:
Infertility affects approximately 1 in 6 couples and may require the use of Medically Assisted Reproduction techniques. In France, there were more than 60,000 in vitro fertilization (IVF) attempts in 2016. The burden of the IVF process is even more significant for working women, causing significant absenteeism due to medical appointments but also to the psychological discomfort caused by the management. Unfortunately, there are no studies that specifically address the quality of life of working women undergoing IVF.

The cohort project aims to measure quality of life using validated questionnaires (FertiQoL, STAI Anxiety Scale and BDI Depression Inventory) in active patients who are scheduled for a first IVF attempt. Quality of life will be measured before starting treatment and at embryo transfer and will be followed up at each embryo transfer for a maximum period of 18 months. The follow-up will end after the live birth of a child or at the end of the 18 months of follow-up.

The investigators will also evaluate, by means of a specific questionnaire, the satisfaction with the interactions between professional and private life (management and consequences of absenteeism at work, consequences on professional evolution, anxious repercussions in the professional and private domains) in the active women undergoing IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Professionally active women aged 18 to 42 years
* Beginning in vitro fertilization treatment at the Montpellier University Hospital

Exclusion Criteria:

* Women who have already had an IVF attempt in the process of egg donation or pre-implantation diagnosis
* History of psychotic or dissociative disorder
* Not fluent in French
* Not affiliated to a social security system
* Protected by law or under curators/guardianship
* No record of non-objection to participate in the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Active women, aged between 18 and 42, undergoing IVF at Montpellier University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the evolution of the quality of life of active patients during their IVF course. | At baseline and through study completion, at 6 months or 12 months or 18 months
  Assessed by the Fertility Quality Of Life (FertiQoL) questionnaire score at 18 months or end of follow-up, compared with the one obtained at inclusion. The score obtained from this questionnaire is not based on a scale.
  2 first items measures physical health and satisfaction with the quality of life in terms of fertility.
  24 other items assesses the impact of fertility problems in several domains: 6 in the emotional, 6 in mind-body, 6 in the relational, 6 in social.
  http://sites.cardiff.ac.uk/fertiqol/description/instrument-description/

SECONDARY OUTCOMES:
Look for predictive factors of impaired quality of life. | At baseline and through study completion, at 6 months or 12 months or 18 months
  Change in the Fertility Quality Of Life (FertiQoL) questionnaire score between baseline and follow-up visits. The score obtained from this questionnaire is not based on a scale.
  2 first items measures physical health and satisfaction with the quality of life in terms of fertility.
  24 other items assesses the impact of fertility problems in several domains: 6 in the emotional, 6 in mind-body, 6 in the relational, 6 in social.
  http://sites.cardiff.ac.uk/fertiqol/description/instrument-description/
Assess work/life interactions and their relationship to quality of life. | At baseline and through study completion, at 6 months or 12 months or 18 months
  Work/life balance satisfaction questionnaire score. This questionnaire consists of 5 questions on the interaction between work and private life. For each question, the patient indicates on a scale from 1 (very unsatisfactory) to 5 (very satisfactory) his level of satisfaction.
Look for predictive factors of dropout. | At baseline and through study completion, at 6 months or 12 months or 18 months
  Anxiety scale score (STAI trait at baseline only, STAI state for all visits). The STAI-Y (State Trait Anxiety Inventory) is a test designed to assess momentary and habitual anxiety.
  The STAI-Y consists of 2 scales of 20 items each:
  * STAY form Y-A (state anxiety): 20 items for how the subject feels in the moment.
  * STAY form Y-B (trait anxiety): 20 propositions to find out what the subject usually feels.
  Each item has a score ranging from 1 to 4 (4 being the highest degree of anxiety). The AE score= sum of the 20 questions on the State page. Ranges from 20 to 80. The AT score= sum of the 20 questions on the Trait page. Varies from 20 to 80.
  Very high: > to 65 High: from 56 to 65 Medium: 46 to 55 Low: 36 to 45 Very low: < or =35
To compare the characteristics of patients who achieve pregnancy versus those who fail (Quality of life, anxiety, depression...) | At baseline and through study completion, at 6 months or 12 months or 18 months
  Beck Depression Inventory (BDI) score. The short validated version is composed of 13 items. This is the most widely used depression questionnaire in the adult population. It provides a quantitative estimate of the intensity of depression. Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity on a scale of 0 to 3.
  The global score of the depressive syndrome (from 0 to 39) is obtained by adding the scores of the 13 items.
  * A score of 0 to 4 corresponds to no depression,
  * From 4 to 7: mild depression,
  * From 8 to 15: moderate depression,
  * A score > 16: severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France